CLINICAL TRIAL: NCT06025591
Title: Role of Ultrasound Elastography in Distinction Between Acute and Chronic Deep Vein Thrombosis: a Prospective Observational Cohort Study
Brief Title: Shear-Wave Elastography in Deep Vein Thrombosis
Acronym: SWE-DVT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Zocco Maria Assunta, Prof, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 5833
Record Dates: First submitted 2023-08-29; First posted 2023-09-06 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Deep Vein Thrombosis
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Compression ultrasonography (CUS), which is the gold-standard for the diagnosis of deep vein thrombosis, cannot provide adequate information on the timing of the onset of thrombosis. Shear-Wave elastography, a technique used to assess tissue elasticity and widely used in hepatology, could play a crucial role in distinguishing between acute and chronic deep vein thrombosis.

This study aims at evaluating the efficacy and diagnostic and prognostic accuracy of Shear-Wave elastography in distinguishing between acute and chronic deep vein thrombosis.

DETAILED DESCRIPTION:
Compression ultrasonography (CUS), supplemented with color-Doppler, is the gold-standard for the diagnosis of deep vein thrombosis. However, it cannot provide adequate information on the timing of the onset of thrombosis, thus not allowing a distinction between acute and chronic venous thrombosis. A few non-standardized and poorly reproducible criteria are used in clinical practice, such as thrombus echogenicity, degree of occlusion and signs of recanalization. The importance of the distinction between acute and chronic venous thrombosis has therapeutic and prognostic implications, especially in patients with occasional and asymptomatic finding of venous thrombosis or in patients with suspected thrombotic recurrence in whom signs and symptoms may be either due to a post-thrombotic syndrome or to a new thrombotic episode.

Shear-Wave elastography, a technique used to assess tissue elasticity and widely used in hepatology, could play a crucial role in distinguishing between acute and chronic deep vein thrombosis. Literature data on the use of this technique in the evaluation of deep venous thrombosis are derived only from observational studies, both retrospective and prospective, mainly based on comparisons between different groups of patients with acute (within 72h from diagnosis) or subacute thrombosis at a 3-months follow-up, with the consequent risk of confounding in the estimating the association of elasticity values to the dating of thrombotic remnant. The few data in the literature on thrombus evolution, assessed by single-patient serialized evaluation, refer to extremely limited case series with short follow-up. In addition, none of these studies consider neoplastic patients, on whom there are no data regarding the usefulness and reproducibility of the method. In accordance with current clinical practice, patients referred to our service of Internal medicine and Thromboembolic Pathology perform ultrasound follow-up so that the evolution of thrombotic residual can be assessed on each patient with large case series and follow-up of longer duration. The primary objective of the present study is to evaluate the efficacy and diagnostic and prognostic accuracy of Shear-Wave elastography in distinguishing between acute and chronic deep vein thrombosis.

Secondary objectives:

* Evaluation of the maximum thickness of the thrombotic residue in compression, as well as the longitudinal extent by B-mode ultrasound method, expressed in mm, at the various time-points of the study
* Evaluation of the degree of venous obstruction, assessed by color-Doppler ultrasound method at the various time-points of the study
* Qualitative evaluation of the echogenicity of the thrombotic remnant, by B-mode ultrasound method in comparison with the echogenicity of the surrounding muscle and vascular structures, at the various time-points of the study.
* Identification of a specific signature for recanalization of deep vein thrombosis of the lower and upper limbs

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* New diagnosis of proximal deep venous thrombosis, Distal deep venous thrombosis of the lower limbs, deep venous thrombosis of the upper limbs, defined as arising within 72 hours prior to the first ultrasound evaluation;
* Availability for follow-up at the above-mentioned Units in Fondazione Policlinico Universitario Agostino Gemelli IRCSS.;
* written informed consent to the participation in the study.

Exclusion Criteria:

* Age <18 years;
* Pregnant or lactating women;
* Life expectancy of less than 6 months;
* Previous performance of drug-mechanical thrombolysis for the treatment of index thrombotic episode;
* Technical impossibility/clinical unreliability of ultrasound evaluation with elastography due to: (a) obligate decubitus of the patient's limb, (b) non-removable occluding dressings, (c) excessive thickness of subcutaneous fatty tissue or edema;
* Previous thrombotic episode at the same site of the thromboembolic episode under study.
* Refusal to sign informed consent to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with newly diagnosed deep venous thrombosis of the lower and upper extremities afferent to the Operating Units of Fondazione Policlinico Universitario Agostino Gemelli IRCSS involved in the study (i.e. Medical Angiology Service, Internal Medicine and Thromboembolic Pathologies and Outpatient Clinic of Internal Medicine and Gastroenterology of the C.E.M.A.D. - Center for Diseases of the Digestive System),who will meet the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Fibrosis Index | 1 month
  Evaluation of a potential time-dependent cut-off of Fibrosis Index discriminating between acute (within 72h) and chronic (3-6-9-12 months) thrombosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Gemelli IRCCS, Roma, Italy